CLINICAL TRIAL: NCT02995486
Title: Effects of a Falls Prevention Program Following Hospital Discharge From a Neuroscience Unit
Brief Title: Effects of a Falls Prevention Program Following Hospital Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: Baptist Health South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-15-0442
Record Dates: First submitted 2016-12-01; First posted 2016-12-16 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Accidental Fall
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Standard care with only an educational pamphlet.
- Intervention (Experimental): Post-discharge exercise group
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Otago Exercise Program for falls prevention after discharge due to fall-related injuries.
  Arms: Intervention

SUMMARY:
A randomized, control trial will be conducted to evaluate the effects of a post-discharge falls prevention program in patients with neurological diseases and disorders. The objective of this study is to evaluate if implementing a falls prevention program is effective in reducing subsequent falls and re-hospitalizations, and improving gait, strength and balance in older adults after hospital discharge. Patients from Baptist Health Neuroscience Center will be randomized on the day of discharge to receive an exercise falls prevention program, delivered by Baptist Health physical therapists, or an educational pamphlet on falls prevention. Baseline and follow up assessments for gait, balance, and strength will be completed at regular intervals to examine effects of the exercise program. In addition, participants will be surveyed to find out about recent falls and hospitalizations. This is a minimal risk study such that the assessments involve conditions in which subjects likely encounter on a daily basis. The risks of the exercise intervention also are no more than one might expect from a community exercise program. Potential benefits include reduced hospitalizations and/or emergency visits related to falls in the intervention group, increased activity levels and improved falls efficacy in the intervention group, and increased system capacity at Baptist Health to deliver a falls prevention program.

DETAILED DESCRIPTION:
After signing the consent form, eligible participants will complete a health-related questionnaire and undergo a gait, balance and strength testing at the time of discharge and then be randomly referred to an intervention (n=30) or to a control group (n=30). Participants will be recruited until the target sample (n=60) is reached. Randomization will be by coin flip.

Measures (intervention and control groups): The evaluation involves non-invasive assessments of physical functioning conducted by physical therapists including balance, gait, and lower limb strength testing. Both groups will be tested by physical therapists at baseline 3, and 6 months post-discharge. A 12-month follow-up call will be made to all participants to ask about falls and physical activity. The physical therapists that conduct the testing will be different from the physical therapists that deliver the intervention (Otago Exercise Program). All tests will be completed in 60-90 minute sessions at Baptist Outpatient Rehabilitation Center. The participants will complete a questionnaire including information on health and falls history, falls self-efficacy (Falls Efficacy Scale), hospitalizations, doctors' visits, and emergency department visits. The participants will also complete a physical assessment including gait analysis using an instrumented mat (GaitRite) to collect data on the temporo-spatial parameters of gait during preferred gait speed and gait during street crossing simulation with regular time: 7 seconds. Street crossing regular time allowance was calculated based on the pre-programmed pedestrian street signals, which give pedestrians 20 seconds to cross a four-lane street. The GaitRite is a thin mat with pressure sensors; an integrated software and web-cam that measures and calculates the gait temporo-spatial parameters. The videos are used only as a visual reference to inspect the task for quality control during data collection and review and will not be used in the analysis or in any other way. The physical assessment will also include the BalanceMaster (Natus Medical, Inc.), a fixed force plate to measure the vertical forces exerted through the feet to measure center of gravity position and postural control, Tinneti Balance Assessment, lower limb strength testing using the 30-second chair stand test, and the Timed Up and Go (TUG) assessment for mobility testing.

Procedures (intervention and control groups): The participants will complete the gait, balance and chair-rise tests in random order. They will be asked a priori to wear non-slip socks provided by the research team. During the preferred gait speed condition, the participants will be instructed to walk on the GAITRite® at their preferred speed as they usually do during their daily activities. During the simulated street crossing condition, the participants will be instructed to cross the street when the pedestrian lights turn green and complete the crossing within the time allowed as displayed by the pedestrian lights on the video. The video includes audio of traffic noise for a more realistic road crossing environment, and it displays an intersection situation in which the subject will be positioned at the intersection, on the sidewalk looking at the oncoming motor vehicle traffic from both directions. A pedestrian light with countdown will also be displayed on the screen. Thus, a functional dual-task paradigm will be used including visual cues and the participants will have to interpret those cues and adjust their gait accordingly. A familiarization trial will be completed, followed by three recording trials under each condition. The order of gait conditions will be randomized for each participant. Participants are free to stop participating at anytime without needing to provide a reason.

Exercise Intervention (intervention group only): The intervention is a comprehensive program addressing aging-related functional decline, fear of falling and inactivity. It targets adults with a history of falls or at-risk for falls. Following the assessments, the participants will be assigned to a control group who will receive the standard educational information on falls prevention, or to an individualized exercise program prescribed and delivered by physical therapists (Otago Exercise Program for Falls Prevention). The program is an easy-to-implement and affordable exercise program for individuals with high risk for falls. The program design model is person-centered and customized to the individual needs. It includes a set of leg muscle strengthening and balance retraining exercises, and a walking plan. Subjects will go to Baptist Outpatient Rehabilitation Center before discharge for the baseline assessment and exercise prescription, then biweekly during the first 2 months (4 times) for exercise progressions and follow ups, once at month 3 for the first re-assessment, then again at 6 months for a booster session and second re-assessment. At 12 months a phone call follow up will be done to ask about falls and physical activity. The assessments and sessions will be covered by the Baptist Health Neuroscience Center and Rehabilitation Services. As part of the program, the participants will do 30 minutes of exercise three times per week, and walk continuously or not for 30 minutes at least two times per week for six months. Participants record (physical activity log) the days they exercise and walk and provide the information to the physical therapists during subsequent visits and/or calls.

Physical therapists will prescribe the exercises based on a large selection available on the program manual. The participants receive an illustration with explanations of the exercises they need to do. They receive a booklet with exercise instructions and ankle cuff weights. The physical therapists will do exercise progressions by increasing intensity and/or difficulty during the subsequent client visits to Baptist Outpatient Rehabilitation Center. The program also includes monthly telephone calls from study staff to maintain motivation, collect information on any falls, and answer questions between visits.

ELIGIBILITY:
Inclusion Criteria:

* Discharged from the hospital after being treated for a fall-related injury;
* Able to engage in an exercise program for falls prevention (sufficient physical and cognitive health);
* Competent to provide consent.

Exclusion Criteria:

* Wheelchair bound;
* Has contraindications for engaging in an exercise program based on the patient records;
* Does not pass the Mini Cog test (brief cognitive screening tool)
* Does not have reliable transportation for follow-up visits.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Self-reported subsequent falls | 12 months

SECONDARY OUTCOMES:
Number of re-hospitalizations | 12 months
Gait velocity in cm/s from a GaitRite instrumented mat | 12 months
Grip strength in N using a Jamar | 12 months
Tinneti Balance Assessment scores | 12 months
Falls Efficacy Scale scores | 12 months
Velocity of center of pressure osculation on the balance master | 12 months
Dorsiflexion strength in N using a hand held dynamometer | 12 months
Step length in cm from a GaitRite instrumented mat | 12 months
Cadence in steps/minute from a GaitRite instrumented mat | 12 months
Step time in seconds from a GaitRite instrumented mat | 12 months
Swing time in seconds from a GaitRite instrumented mat | 12 months
Stance time in seconds from a GaitRite instrumented mat | 12 months
Double-support time in seconds from a GaitRite instrumented mat | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Edgar R Vieira, Principal Investigator — Florida International University
Locations (1):
- Baptist Hospital, Miami, Florida, United States